CLINICAL TRIAL: NCT04932668
Title: The Feasibility and Impact of A Home-Based NMES Program on Post-Stroke Lower Limb Spasticity
Brief Title: Home Based Electrical Stimulation on Post-stroke Lower Limb Tightness.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Raja Nabila binti Raja Mohamed Anuar, Doctor, Principal Investigator, University of Malaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020427-8560
Record Dates: First submitted 2021-06-06; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Spasticity as Sequela of Stroke

STUDY DESIGN:
Intervention Model Description: To evaluate the feasibility and acceptability of a home-based NMES program on lower limb spasticity in patient with post-stroke
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based Electrical Stimulation Program for lower limb spasticity (Experimental): Single arm prospective intervention study to assess the feasibility and impact of a home-based program. Patient will apply home-based NMES on their leg for 20 minutes, 5 days a week for 4 weeks. At the end of the study, an outcome measures will be assessed and patient will be required to answer a questionnaires on their experience.
  Interventions: Other: Feasibility and Impact of Home-based Electrical Stimulation Program

INTERVENTIONS:
Other: Feasibility and Impact of Home-based Electrical Stimulation Program — Home-based NMES program on spastic leg. The NMES pre-programmed dosage (locked):
  NMES waveform is biphasic PC, Frequency 50Hz, pulse width 400µs, ON:OFF 10s:20s and current amplitude: individual maximum tolerated to achieve ankle dorsiflexion.
  Other Names: Program

SUMMARY:
Spasticity is a common complication post stroke. Post-stroke spasticity along with weakness and lack of coordination result in gait abnormalities and functional limitations. Recent treatment option include neuromuscular electric stimulation (NMES), a form of therapy that applies electrical currents to produce contraction of innervated muscle by depolarizing local motor nerves. Currently, there are wide varieties of NMES devices available commercially for consumer.

The main purpose of this study is to evaluate the feasibility and acceptability of a home-based NMES program on lower limb spasticity in patient with post-stroke more than 6 months and to assess the impact of the program. This is single arm prospective intervention study. Patient will apply home-based NMES on their leg for 20 minutes, 5 days a week for 4 weeks. At the end of the study, an outcome measures will be assessed and patient will be required to answer a questionnaires on their experience.

ELIGIBILITY:
Inclusion Criteria:

1. Post stroke (hemorrhagic or ischemic) with ankle plantarflexor (gastrocnemius and soleus) spasticity MAS 1+ to MAS 3,
2. Post stroke more than 6 months,
3. At least 18 years old,
4. Able to ambulate 10 meter either independently or aided (single point stick or quadripod)
5. Compliant to outpatient therapy.
6. Minimal cognitive (MMSE> 24) and minimal sensory impairment,
7. Stable neurological and medical condition

Exclusion Criteria:

1. Introduction or changes in anti-spastic medication dose within 3 months or during study period,
2. Receiving intervention for spasticity (eg BoNT or serial casting) within 3 months or during research period,
3. New neurological condition/disease,
4. Presence of contraindications to NMES, which is: Pregnancy, Malignancy, Presence of electronic implant eg cardiac pacemaker, cardioverter defibrillator, Uncontrolled seizure/epilepsy, Infected tissues/ tuberculosis or osteomyelitis, Impaired lower limb circulation/ DVT/ thrombophlebitis, Recent fracture or osteoporosis, Actively bleeding tissue or person with untreated hemorrhagic disorder, Damaged or skin diseases at the affected lower limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Retention Rate | 4 weeks
  The proportion of patients who completed the program. Patient completed divided with patient recruited, expressed in percentage (%).
Acceptability | 4 weeks
  Acceptability as evaluated at the end of the intervention by brief structured questionnaire developed for this study using 5 point Likert scale with 1 (strongly agree) and 5 (strongly agree).

SECONDARY OUTCOMES:
Clinical measurement of spasticity | 4 weeks (pre and post assessment)
  Ankle dorsiflexor (gastroc) Modified Ashworth Scale (MAS) as measured in MAS grade 1, 1+, 2, 3, 4
Clinical measurement of spasticity | 4 weeks (pre and post assessment)
  Modified Tardieu Scale (R1 and R2 angle of ankle dorsiflexion)
Ankle dorsiflexion muscle strength | 4 weeks (pre and post assessment)
  Manual Muscle Testing as measured in 0-5 (with 0 no movement and 5 is the strongest)
Functional Outcome | 4 weeks (pre and post assessment)
  10 meter walking test

CONTACTS AND LOCATIONS:
Overall Officials: Raja Nabila BT Raja Mohamed Anuar, Principal Investigator — University Malaya Medical Center
Locations (1):
- University Malaya Medical Center, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT04932668/Prot_000.pdf
  • Informed Consent Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT04932668/ICF_001.pdf